CLINICAL TRIAL: NCT06679049
Title: Comparison of Healing Measures in Diaphyseal Tibial Fractures Following Standard Intramedullary Nailing or Micromotion Tibial Intramedullary Nailing
Brief Title: Comparison of Healing Measures Tibial Fractures Following Standard Intramedullary Nailing or Micromotion Tibial Intramedullary Nailing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Joseph Johnson, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 300013319; UAB (Other: UAB)
Record Dates: First submitted 2024-11-06; First posted 2024-11-07 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Tibial Fractures
MeSH Terms: conditions — Tibial Fractures

STUDY DESIGN:
Intervention Model Description: Subjects Undergoing Tibial Fracture Repair
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Micromotion Cohort (Experimental): use of at least 2 distal interlocking screws and the use of a minimum of 1 proximal tibial interlocking screw
  Interventions: Procedure: micromotion intramedullary nail cohort
- Standard Cohort (Experimental): use of at least 2 distal interlocking screws and the use of a minimum of 1 proximal interlocking screw
  Interventions: Procedure: standard intramedullary nail cohort

INTERVENTIONS:
Procedure: micromotion intramedullary nail cohort — use of at least 2 distal interlocking screws and the use of a minimum of 1 proximal tibial interlocking screw
  Arms: Micromotion Cohort
Procedure: standard intramedullary nail cohort — use of at least 2 distal interlocking screws and the use of a minimum of 1 proximal interlocking screw
  Arms: Standard Cohort

SUMMARY:
The primary purpose of this study is to perform a high-quality randomized control trial comparing intramedullary tibial nail fixation with standard design nails to a micromotion tibial nail device, to evaluate the rates of union and post-operative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 85 years
* Stable Tibial fracture recommended for surgical intervention

Exclusion Criteria:

* Patients not meeting inclusion criteria
* Unstable fracture patterns e.g. those needing a secondary intervention - masquelet/cement spacer)
* Previously non-ambulatory patients
* Delayed presentation of fracture (>4 weeks)
* Fractures that the treating surgeon indicates requires additional fixation strategies to achieve stability
* Patients with an achieve infection or wound at the surgical site
* Any previous ligament or fracture surgery on the index site
* Inflammatory rheumatic disease or other rheumatic disease-
* Immune compromised patients (hepatitis, HIV, etc.)
* Unwilling or unable to participate or follow study protocol

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
The difference in radiographic union | 12,18 and 24 weeks between micromotion intramedullary fixation and standard IMN post operatively
  bridging callus, minimum three cortices bridged

SECONDARY OUTCOMES:
difference in complication rates | 1 year post-operatively
  Patient reported outcomes scores

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Johnson, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham Main Hospital, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No